CLINICAL TRIAL: NCT03645239
Title: Post-operative Emesis and Pain Outcomes After Cesarean Delivery (EPOC)
Brief Title: Post-operative Emesis and Pain Outcomes After Cesarean Delivery
Acronym: EPOC
Status: Active, not recruiting | Type: Observational
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANAESPRG18/02
Record Dates: First submitted 2018-08-05; First posted 2018-08-24 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Pain, Postoperative; Cesarean Section; Nausea, Postoperative; Vomiting, Postoperative
Keywords: Postoperative pain; Cesarean delivery; Postoperative nausea and vomiting
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control: Questionnaires, Mechanical Temporal Summation assessment and preoperative pain assessment will be assigned to patient. Patients will be assigned to this group when they have a pain score of less than 3 (out of 10) at 6-10 post-delivery online/phone survey.
  Interventions: Procedure: Mechanical Temporal Summation assessment; Other: Preoperative pain assessment; Other: Questionnaires
- Postoperative pain: Questionnaires, Mechanical Temporal Summation assessment and preoperative pain assessment will be assigned to patient. Patients will be assigned to this group when they have a pain score of equal or more than 3 (out of 10) at 6-10 post-delivery online/phone survey.
  Interventions: Procedure: Mechanical Temporal Summation assessment; Other: Preoperative pain assessment; Other: Questionnaires
- Control (non-Headspace): Questionnaires, Mechanical Temporal Summation assessment and preoperative pain assessment will be assigned to patient. Twenty five patients will be assigned to this group when they agree to participate in a sub-study on the use of a mindfulness exercise mobile app (Headspace). Patients will have a follow-up online/phone call survey at day 7-20 and 4-8 weeks after delivery.
  Interventions: Procedure: Mechanical Temporal Summation assessment; Other: Preoperative pain assessment; Other: Questionnaires
- Experimental (Headspace): Questionnaires, Mechanical Temporal Summation assessment and preoperative pain assessment will be assigned to patient. Fifty five patients will be assigned to this group when they agree to participate in a sub-study on the use of a mindfulness exercise mobile app (Headspace). Patients will have a follow-up online/phone call survey at day 7-20 and 4-8 weeks after delivery.
  Interventions: Procedure: Mechanical Temporal Summation assessment; Other: Preoperative pain assessment; Other: Questionnaires; Other: Headspace

INTERVENTIONS:
Procedure: Mechanical Temporal Summation assessment — A 180 gram von Frey filament is applied on the subject's forearm. Patient will then be asked to rate the pinprick pain score on a verbal rating scale, 0-100. Following this, 10 consecutive touches at random locations are applied with a 1 second interstimulus interval and within a 1 cm diameter circle. The patient will then be asked to rate the 10th pain score (0-100). The Mechanical Temporal Summation Score is obtained by the difference between the 11th pain score and the 1st pain score. If the score is greater than zero, the patient is implied to have presence of Mechanical Temporal Summation.
  Other Names: MTS
Other: Preoperative pain assessment — Patients will be asked to rate, using a 0-10mm visual analog scale (VAS), their surgical anxiety level ("On a scale of 0-100, with 0 being not anxious at all to 100 being extremely anxious, how anxious are you about your upcoming surgery?"), their anticipated pain (On a scale of 0-10, with 0 being no pain at all and 10 being pain as bad as you can imagine, how much pain do you anticipate experiencing after your upcoming surgery?"), and using a categorical scale, their anticipated pain medication need ("On a scale of 0 to 5, with 0 being none at all, 1 being much less than average, 2 being less than average, 3 being average, 4 being more than average, and 5 being much more than average, how much pain medication do you anticipate needing after your upcoming surgery?").
Other: Questionnaires — Questionnaires including Hospital Anxiety and Depression Scale (HADS), EQ-5D-3L, Edinburgh Postnatal Depression Scale (EPDS), Pain Catastrophizing Scale (PCS), Central Sensitisation Inventory (CSI), pain survey and breastfeeding questionnaire will be administered to the patient.
Other: Headspace — The mindfulness exercise mobile application, Headspace, will be downloaded into the patients' mobile devices. Patients will be asked to experience a mindfulness exercise for 10-30 minutes before delivery. HADS and pain score will be asked after the intervention.
  Groups: Experimental (Headspace)

SUMMARY:
Approximately 20% women who undergo cesarean delivery would suffer from severe post-operative pain, which may further increase their risks from developing postpartum depression. Predictive factors such as pre-operative pain, age and anxiety could significantly contribute to post-operative nausea and vomiting (PONV) and pain in general surgery, however little information is available with regards to cesarean delivery. The investigators would investigate the risk factors of causing post-operative emesis after cesarean delivery, and to reaffirm that there is a positive correlation between pain on local anesthetic injection, presence of mechanical temporal summation (MTS) and post-Cesarean pain scores.

DETAILED DESCRIPTION:
Previous studies demonstrated that pain scores upon local anesthetic injection is positively correlated to post-cesarean pain scores. Anxiety, anticipated post-operative pain score and anticipated medication need are also found to be promising risk factors to post-cesarean pain management.

The investigators would investigate the risk factors of causing post-cesarean emesis, and to reaffirm that there is a positive correlation between pain on local anesthetic injection, presence of mechanical temporal summation (MTS) and post-Cesarean pain scores. 470 parturients undergoing cesarean delivery and requiring regional anaesthesia will be recruited. Pain and anxiety assessment will be conducted via visual analogue scoring (VAS), MTS assessment and a series of questionnaires. After delivery, patients will be given appropriate analgesia, and pain score at movement will be recorded. Secondary outcomes include pain scores at rest, analgesia consumption, time-to-first-rescue analgesia, opioid-related side effects, patient satisfaction and postpartum depression. A separate 125 patients will be recruited to evaluate the feasibility and patient acceptability of the use of Headspace, a mindfulness mobile application during the pre- and postnatal period to improve the maternal outcomes (emesis, pain, anxiety, depression).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant and going to have caesarean delivery (36 weeks gestation or more; nulliparous and multiparous);
* Healthy or have mild medical problems that are well-controlled (American Society of Anesthesiologists physical status 1-2).

Exclusion Criteria:

* History of intravenous drug or opioid abuse;
* Previous history of chronic pain syndrome;
* Emergency cesarean section;
* Undergo general anaesthesia during cesarean delivery;
* Non-English speaking.

Ages: 21 Years to 50 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Only female undergoing cesarean delivery in the institution will be recruited.
Study Population: Pregnant females undergoing cesarean delivery.
Sampling Method: Non-Probability Sample
Enrollment: 595 (Estimated)
Dates: Start 2018-05-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Postsurgical pain scores in both groups: Numeric Rating Scale | 6 -10 weeks after delivery
  Pain scores (Numeric Rating Scale 0-10) at 6-10 weeks follow-up evaluations. Zero being no pain, and 10 being the worst pain possible.

SECONDARY OUTCOMES:
Pain vulnerability in both groups: Pain Catastrophizing Scale | 7 weeks (Upon recruitment until 5-14 days after delivery)
  Assessment will be done via Pain Catastrophizing Scale (PCS) questionnaire before surgery. Pain catastrophizing refers to the negative thought processes patients have when they are exposed to pain or painful experiences. The PCS is a 13-item scale, with each item rated on a 5-point scale: 0 (Not at all) to 4 (all the time). It is broken into three subscales being magnification (0-12), rumination (0-16), and helplessness (0-24). A higher value in each subscale indicates a higher tendency to that subscale (worse outcome).
Mechanical Temporal Summation as measured by von Frey filament in both groups | 1 day (10 minutes)
  Assessment will be done via Mechanical Temporal Summation assessment before surgery. A 180 gram von Frey filament is applied on the subject's forearm. Patient will then be asked to rate the pinprick pain score on a verbal rating scale, 0-100. Following this, 10 consecutive touches at random locations are applied with a 1 second interstimulus interval and within a 1 cm diameter circle. The patient will then be asked to rate the 10th pain score (0-100). The Mechanical Temporal Summation Score is obtained by the difference between the 11th pain score and the 1st pain score. If the score is greater than zero, the patient is implied to have presence of Mechanical Temporal Summation.
Edinburgh Postnatal Depression Scale (EPDS) before and after delivery | 6 -10 weeks after delivery
  Edinburgh Postnatal Depression Scale (EPDS) is a 10-item self reporting scale to evaluate the postnatal depression. Participants are asked to respond according to how they have felt in the past seven days. Each item is measured on a 4-point scale (0-3), with a total score in the range of 0 to 30. A higher total score indicates a greater degree of depressive symptoms. A score of 10 and above indicates clinically significant depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Farida Ithnin, MB BCh BAO, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tan HS, Tan CW, Sultana R, Lim CH, Chan JJI, Habib AS, Sng BL. Factors associated with postoperative nausea or vomiting in parturients undergoing caesarean delivery under spinal anaesthesia with intrathecal morphine: A prospective cohort study. Eur J Anaesthesiol. 2022 Jan 1;39(1):75-77. doi: 10.1097/EJA.0000000000001427. No abstract available. PMID 34857684

DOCUMENTS (1):
  • Study Protocol (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT03645239/Prot_000.pdf